CLINICAL TRIAL: NCT00237978
Title: Control of Therapy of Acne Papulopustulosa by Visible Light With Waterfiltered Infrared and / or Adapalen (Differin Gel)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Roland Aschoff, MD, Technical University Dresden
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TUD-Akne02-003
Record Dates: First submitted 2005-10-12; First posted 2005-10-13 (Estimated); Last update posted 2009-05-14 (Estimated); Status verified 2008-05

CONDITIONS: Acne Papulopustulosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): VIS and wIRA
  Interventions: Radiation: VIS and wIRA
- 2 (Active Comparator): VIS, wIRA and Adapalen
  Interventions: Drug: Adapalen; Radiation: VIS and wIRA
- 3 (Active Comparator): Adapalen
  Interventions: Drug: Adapalen

INTERVENTIONS:
Drug: Adapalen
  Arms: 2; 3
Radiation: VIS and wIRA
  Arms: 1; 2

SUMMARY:
The aim of the study is to investigate the effectivity of visible light in combination with waterfiltered infrared in treating acne papulopustulosa. The reduction of inflammatory and non-inflammatory lesions within 8 weeks will be measured and compared with the standard treatment with Adapalene.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate acne papulopustulosa according to Burton Scale Stage 3 to 4
* At least 5 inflammatory and 5 non-inflammatory lesions in the face
* Age >= 14 years

Exclusion Criteria:

* pregnant and nursing women
* Antiandrogen therapy
* therapy with antibiotics within the last 4 weeks
* therapy with retinoids within the last 6 months
* natural or artificial UV-therapy within the last 4 weeks
* severe acne papulopustulosa according to Burton Scale 5 or 6
* Severe systemic condition
* Secondary acne

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-09; Primary Completion 2009-06 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
reduction of inflammatory and non-inflammatory lesions within 8 weeks after start of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Roland Aschoff, MD, Principal Investigator — Technische Universität Dresden, Fetscher Str. 74, 01307 Dresden, Germany
Locations (1):
- Universitätsklinikum Carl Gustav Carus an der Technischen Universität Dresden, Dresden, Saxony, Germany